CLINICAL TRIAL: NCT01039493
Title: Living With Cervical Cancer: Assessing Utilities Associated With Common Treatment Complications
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2009-1240; OS09708 (Other: UW Carbone Cancer Center)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients
- Providers

SUMMARY:
The objective of this study is to establish patient preferences in regards to common complications of cervical cancer treatments, and to compare these preferences to those of medical providers who care for cervical cancer patients. These preferences will be determined via a interview using the Standard Gamble, which is a well-recognized method for establishing utilities.

ELIGIBILITY:
Inclusion Criteria:

* A subject has to have been diagnosed with early cervical cancer (Stage I or II) within the last 3 years and/or take care of patients with cervical cancer and identify her or himself as one of the following: gynecologic oncologist, radiation oncologist, physician's assistant or nurse.
* Subjects must be ≥18 and <61 years old.

Exclusion Criteria:

* Subjects who are unable to read and speak English proficiently will be excluded. Proficiency will be assessed by the investigator enrolling patients.
* Subjects who do not have capacity to consent will not be included in this study.
* Subjects may not be investigators on this study.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient Population: Patients ≥18 and <61 years old who were diagnosed with early cervical cancer (stages I and II) at least 3 years prior to the interview. We cannot limit our population to stage IB2 patients and meet our accrual goals due to the rarity of the disease. Patients with stages I and II cervical cancer are included because they have the potential to be exposed to the same treatment complications as patients with stage IB2 disease. Patients of all health statuses will be accepted.
  Provider Population: Providers who care for patients with cervical cancer at the University of Wisconsin, including: gynecologic oncologists, radiation oncologists, physician's assistants and nurses. Providers must be ≥18 and <61 years old in any health status.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Utilities of complications associated with cervical cancer treatment. | At time of interview

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Hartenbach, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States